CLINICAL TRIAL: NCT01509807
Title: A Pain Relief Trial Utilizing the Infiltration of a Multivesicular Liposome Formulation Of BupiVacaine, EXPAREL®: A Phase 4 Health Economic Trial in Adult Patients Undergoing Ileostomy Reversal
Brief Title: A Health Economic Trial in Adult Patients Undergoing Ileostomy Reversal MA402S23B504
Acronym: IMPROVE-IR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Collaborators: Registrat-Mapi (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MA402S23B504
Record Dates: First submitted 2011-10-24; First posted 2012-01-13 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-03

CONDITIONS: Retraction of Colostomy
Keywords: Ileostomy reversal
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): IV morphine sulfate (or Sponsor-approved equivalent), Standard of Care (SOC)
  Interventions: Drug: IV morphine sulfate or Sponsor-approved equivalent
- Group 2 (Experimental): EXPAREL (bupivacaine liposome injectable suspension)
  Interventions: Drug: EXPAREL

INTERVENTIONS:
Drug: IV morphine sulfate or Sponsor-approved equivalent — Patients enrolled in this group will receive IV morphine sulfate or Sponsor-approved equivalent via a patient-controlled analgesia (PCA) pump, as needed.
  Arms: Group 1
Drug: EXPAREL — Patients enrolled in this group will receive 266 mg EXPAREL diluted with preservative-free 0.9% normal saline to a total volume of 30 cc and administered via wound infiltration prior to wound closure. When not contraindicated, 30 mg IV ketorolac will be given at the end of surgery. If not indicated, IV non-steroidal anti-inflammatory drug (NSAID) may be substituted per the site's standard of care.
  Other Names: bupivacaine liposome injectable suspension
  Arms: Group 2

SUMMARY:
This study is designed to compare the standard of care against EXPAREL (bupivacaine liposome injectable suspension) to determine if total opioid consumption is reduced when using EXPAREL, therefore possibly reducing total hospitalization costs.

DETAILED DESCRIPTION:
This is a phase 4, prospective, sequential, open-label study designed to evaluate the efficacy, safety, and health economic benefits of intraoperative local wound infiltration with EXPAREL (bupivacaine liposome injectable suspension) compared with postsurgical administration of standardized intravenous (IV) morphine sulfate for postsurgical analgesia in adult patients undergoing ileostomy reversal with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age and older
* Patients scheduled to undergo ileostomy reversal
* Ability to provide informed consent, adhere to study visit schedule, and complete all assessments.

Exclusion Criteria:

* Patients with a history of hypersensitivity or idiosyncratic reactions or intolerance to any local anesthetic, opioid, or propofol.
* Patients who abuse alcohol or other drug substance.
* Patients with severe hepatic impairment.
* Patients currently pregnant or who may become pregnant during the course of the study or who are unwilling to use acceptable means of contraception for at lest one month before and one month after dosing.
* Patients with any psychiatric, psychological, or other condition that the Investigator feels may make the patient an inappropriate candidate for this clinical study.
* Patients who have participated in an EXPAREL study within the last 30 days.
* Patients who have received an investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during the patient's participation in this study.

In addition, the patient will be ineligible if he/she meets the following criteria during surgery:

* Patients who have any concurrent surgical procedure.
* Patients who receive intraoperative administration of opioids (other than fentanyl or analogs) or any other analgesic, local anesthetics, or anti-inflammatory agents.
* Patients who receive Entereg(R).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Marcet, MD, Principal Investigator — University of South Florida, Tampa, FL; Valentine Nfonsam, MD, Principal Investigator — University of Arizona, Tucson, AZ; Sergio Larach, MD, Principal Investigator — Florida Hospital, Orlando, FL.
Locations (3):
- United States (3):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Florida Hospital d/b/a Colon & Rectal Surgery Center, Orlando, Florida
  - University of South Florida, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 16 | 17
Completed | 15 | 16
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: One patient in Group 1 did not have the planned surgery. Thus, while 16 participants were enrolled in Group 1, 15 participants were in the Safety Analysis Set and had the planned surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (16.03) | 52.1 (15.89) | 53.8 (15.8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Burden
Description: Total opioid consumed (IV and PO) postsurgically until hospital discharge order is written or through Day 30, whichever is sooner.
Time Frame: Wound closure to time the discharge order is written or Day 30, whichever is sooner
Population: The Efficacy Analysis Set had 11 participants in Group 1 and 16 participants in Group 2. The Efficacy Analysis Set was defined as those patients who underwent the planned surgery, did not meet any of the intraoperative exclusion criteria, and had provided informed consent. In addition, the Group 2 patients must have received study drug (EXPAREL).
Measure: Mean (Standard Deviation); unit: mg morphine equivalent
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 16
mg morphine equivalent | 112.38 (117.08) | 19.8 (34.08)

2. Primary Outcome: Health Economic Benefits - Total Cost of Hospitalization
Description: 1) Total cost of hospitalization until the time hospital discharge order is written or through Day 30, whichever is sooner.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 16
dollars | 9950.47 (3899.04) | 6728.88 (1874.89)

3. Secondary Outcome: Incidence of Opioid-related Adverse Events
Description: Incidence of opioid-related adverse events defined as somnolence, respiratory depression, hypoventilation, hypoxia, dry mouth, nausea, vomiting, constipation, sedation, confusion, pruritus, urinary retention, and postoperative ileus.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 16
events | 6 (0.82) | 4 (0.45)

4. Primary Outcome: Health Economic Benefit - Length of Stay
Description: Time from completion of wound closure until hospital discharge written or through Day 30, whichever was sooner
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 16
days | 5.1 [2.2 to 31.9] | 3 [0.8 to 5]

5. Secondary Outcome: Patient Satisfaction With Postsurgical Analgesia
Description: Responses to question pertaining to patient satisfaction with postsurgical analgesia described by total percentage indicating satisfied or extremely satisfied.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 16
percentage of patients | 90.91 (0.65) | 87.5 (0.83)

6. Secondary Outcome: Patient Discharged From the Hospital for at Least 3 Days
Description: Yes, if patient was discharged from the hospital for at least 3 days; no, if patient was not discharged for at least 3 day; not reported if appropriate
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 16
participants | 11 | 14

7. Secondary Outcome: Readmission to Hospital Since Discharge
Description: Yes, if patient was readmitted to hospital since discharge; no, if patient was not readmitted to hospital since discharge; not reported, if appropriate.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 16
participants | 0 | 0

8. Secondary Outcome: Make Unplanned VIsit(s) With Any Healthcare Providers
Description: Yes, if patient made an unplanned visit with a healthcare provider; no, if patient did not make an unplanned visit with a healthcare provider; not reported, if applicable
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 16
participants | 1 | 0

9. Secondary Outcome: Contact or Attempt to Contact Surgeon/Doctor to Discuss Recovery After Surgery
Description: Yes, if patient contacted or attempted to contact surgeon/doctor to discuss recovery after surgery; no, if patient did not contact or attempt contact; not reported if applicable.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 16
participants | 1 | 0

10. Secondary Outcome: Experienced Any Health Problems or Changed in Health Since Hospital Discharge
Description: Yes, if patient experienced any health problems or changes in health since hospital discharge; no, if patient did not experience health problems or changes since hospital discharge; not reported, if applicable.
Time Frame: Wound closure to time hospital discharge order is written or Day 30, whichever is sooner.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 11 | 16
participants | 1 | 2

ADVERSE EVENTS:
Description: The Safety Analysis Set included all patients who underwent the planned surgery. There were 15 participants in Group 1 and 17 participants in Group 2 who underwent the planned surgery.
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/17
Other Adverse Events (participants affected / at risk) | 7/15 | 8/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=15) | Group 2 (N=17)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=15) | Group 2 (N=17)
Abdominal distention (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 3 (3) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Anal injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site edema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Incisional drainage (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No